CLINICAL TRIAL: NCT02647281
Title: A Double-Blind, Placebo-Controlled, Dose-Escalation, First Time in Human Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of GSK3389404 in Healthy Subjects
Brief Title: First Time in Human Study to Assess the Safety, Tolerability and Pharmacokinetics of GSK3389404 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 202007; 2015-003781-84 (EudraCT Number)
Record Dates: First submitted 2015-12-14; First posted 2016-01-06 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Hepatitis B
Keywords: Single dose; Multiple ascending doses (MAD); Pharmacokinetics; Safety; GSK3389404; Tolerability
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Part 1: GSK3389404 10 mg (Experimental): Subjects will receive a single dose of GSK3389404 10 mg by subcutaneous injection on Day 1 of Part 1.
  Interventions: Drug: GSK3389404
- Part 1: Placebo (Placebo Comparator): Subjects will receive a single dose of subcutaneous (injection under the skin) injection of placebo matching with GSK3389404 10 milligram (mg) or 30 mg, or 60 mg or 120 mg.
  Interventions: Drug: Matching Placebo
- Part 1: GSK3389404 30 mg (Experimental): Subjects will receive a single dose of GSK3389404 30 mg by subcutaneous injection on Day 1 of Part 1.
  Interventions: Drug: GSK3389404
- Part 1: GSK3389404 60 mg (Experimental): Subjects will receive a single dose of GSK3389404 60 mg by subcutaneous injection on Day 1 of Part 1.
  Interventions: Drug: GSK3389404
- Part 1: GSK3389404 120 mg (Experimental): Subjects will receive a single dose of GSK3389404 120 mg by subcutaneous injection on Day 1 of Part 1.
  Interventions: Drug: GSK3389404
- Part 2: GSK3389404 30 mg (Experimental): Subjects will receive a single dose of GSK3389404 30 mg by subcutaneous injection QW for 4 weeks in Part 2.
  Interventions: Drug: GSK3389404
- Part 2: Placebo (Placebo Comparator): Subjects will receive a single dose of subcutaneous injection of placebo matching with GSK3389404 30 mg or 60 mg or 120 mg once weekly (QW) for 4 weeks in Part 2.
  Interventions: Drug: Matching Placebo
- Part 2: GSK3389404 60 mg (Experimental): Subjects will receive a single dose of GSK3389404 60 mg by subcutaneous injection QW for 4 weeks in Part 2.
  Interventions: Drug: GSK3389404
- Part 2: GSK3389404 120 mg (Experimental): Subjects will receive a single dose of GSK3389404 120 mg by subcutaneous injection QW for 4 weeks in Part 2.
  Interventions: Drug: GSK3389404

INTERVENTIONS:
Drug: GSK3389404 — GSK3389404 is supplied as solution for injection vial. Each vial contains 100 mg/mL of GSK3389404. It's physical appearance is clear colourless to slightly yellow solution.
  Arms: Part 1: GSK3389404 10 mg; Part 1: GSK3389404 120 mg; Part 1: GSK3389404 30 mg; Part 1: GSK3389404 60 mg; Part 2: GSK3389404 120 mg; Part 2: GSK3389404 30 mg; Part 2: GSK3389404 60 mg
Drug: Matching Placebo — Placebo is supplied as solution for injection vial. It's physical appearance is clear colourless solution.
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
This study is a Phase 1, randomized, double-blind (Sponsor unblinded), placebo controlled, dose escalation study to determine the safety, tolerability and pharmacokinetics (PK) profile of GSK3389404 as single (Part 1) and multiple subcutaneous (SC) injections (Part 2) in healthy subjects. This study represents the first administration of GSK3389404 in humans to define the safety, tolerability and PK following single and multiple doses of GSK3389404 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions and is likely to complete the study as planned.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and electrocardiograms (ECGs). There should be no evidence of cardiac, pulmonary, hepatic, biliary, gastrointestinal, or renal disorders, or cancer within the past 5 years (except localized or in situ cancer of the skin). A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria and are reported as outside of the normal reference range for healthy subjects may be included only if the Investigator considers the finding unlikely to introduce additional risk to the subject and will not interfere with the study procedures.
* Male or female between 18 and 55 years of age, inclusive, at the time of signing the informed consent form (ICF).
* Body weight >50 kilograms (kg) (110 pounds [lb]) for men and >45 kg (99 lb) women and a body mass index (BMI) between 18 to 30 kg/meter-squared, inclusive, will be allowed.
* AST, ALT, ALP, bilirubin, and creatinine within the normal reference range. If outside the normal reference range, these values may be repeated once at the discretion of the Investigator or designee.
* WBC count (including neutrophil counts), haemoglobin and platelets within the normal reference range. If outside the normal reference range, these values may be repeated once at the discretion of the Investigator or designee.
* Females of Reproductive Potential (FRP) are not permitted. Eligible females must meet the following criteria:

  * Non-pregnant (as confirmed by a negative serum human chorionic gonadotrophin (hCG) test); AND
  * Non-lactating at screening and prior to dosing; AND
  * Non-reproductive potential as defined by at least one of the following conditions: Pre-menopausal females without reproductive potential defined by one of the following: Documented salpingectomy, Hysterectomy, Documented bilateral oophorectomy; Postmenopausal defined as 12 months of spontaneous amenorrhea; A blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels may be conducted at the discretion of the Investigator or site to confirm non-reproductive potential.
* Male subjects with female partners of child-bearing potential must agree to meet one of the contraception requirements from the time of first dose of study treatment until the last follow-up visit (Part 1 Day 60; Part 2 Day 113).

  * Vasectomy with documentation of azoospermia.
  * Male condom plus partner use of one of the contraceptive options below that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label: Contraceptive subdermal implant; Intrauterine device or intrauterine system; Combined estrogen and progestogen oral contraceptive; Injectable progestogen; Contraceptive vaginal ring; Percutaneous contraceptive patches These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The Investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

Exclusion Criteria:

* History or other clinical evidence of hypertension, significant or unstable cardiac disease (e.g., prolonged QT syndrome [torsade de pointes], angina, congestive heart failure, myocardial infarction, diastolic dysfunction, significant arrhythmia, coronary heart disease and/or clinically significant ECG abnormalities).
* History of, or active diagnosis of, liver disease such as Gilbert's syndrome, cirrhosis, autoimmune hepatitis, non-alcoholic fatty liver disease /non-alcoholic steatohepatitis, or hemochromatosis.
* History of, or active diagnosis of, primary or secondary (e.g., renal disease secondary to diabetes, hypertension, vascular disease, etc.) renal disease.
* History of bleeding diathesis or coagulopathy.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 milliliters [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Unwilling to abstain from alcohol for 48 hours prior to the start of dosing until the last dose in each dosing session.
* Regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* History of sensitivity to GSK3389404 or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including vitamin, dietary and herbal supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study treatment.
* Use of aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) within 7 days prior to the first dose of study treatment.
* A positive hepatitis C antibody.
* A positive pre-study Hepatitis B surface antigen (HBsAg).
* A positive test for human immunodeficiency virus (HIV) antibody.
* Serum creatinine greater than the upper limit of normal (ULN)
* Glomerular filtration rate <90 mL/minute as calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-epi) formula
* Albumin to creatinine ratio (ACR) >= 0.03 milligram/milligram (mg/mg). In the event of an ACR above this threshold, eligibility may be confirmed by a second measurement.
* Qualitative test (urinalysis) for blood in urine >= 0.03 mg/deciliter. In the event of a positive test, the test may be repeated once, and if negative, the subject considered eligible.
* A positive pre-study drug screen. Unwilling to refrain from use of the illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* Fridericia's QT correction formula (QTcF) >= 450 milliseconds (msec).
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 5 half-lives (if known) or twice the duration (if known) of the biological effect of the study drug (whichever is longer) or 90 days (if half-life or duration is unknown).
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Prior treatment with any oligonucleotide or small interfering ribonucleic acid (siRNA) within 12 months prior to the first dosing day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=202007

REFERENCES:
- [Background] Han K, Cremer J, Elston R, Oliver S, Baptiste-Brown S, Chen S, Gardiner D, Davies M, Saunders J, Hamatake R, Losos J, Leivers M, Hood S, van der Berg F, Paff M, Ritter JM, Theodore D. A Randomized, Double-Blind, Placebo-Controlled, First-Time-in-Human Study to Assess the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of GSK3389404 in Healthy Subjects. Clin Pharmacol Drug Dev. 2019 Aug;8(6):790-801. doi: 10.1002/cpdd.670. Epub 2019 Mar 12. PMID 30861337

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 1, randomized, double-blind (sponsor un-blinded), placebo-controlled, dose escalation study to determine the safety, tolerability, and pharmacokinetic (PK) profile of GSK3389404 as single and multiple subcutaneous (SC) injections in healthy participants. This study was conducted at 2 centers in London, United Kingdom.
Pre-assignment Details: The study was conducted in 2 Parts: Single-Ascending Dose (Part 1) and Multiple-Ascending Dose (Part 2). In Part 1, total of 32 participants were enrolled and all of them were randomized to receive the study treatment. In Part 2, a total of 24 participants were enrolled and all of them were randomized to receive the study treatment.
Groups:
- Part 1: Placebo: Participant received a single dose of subcutaneous (injection under the skin) injection of placebo matching with GSK3389404 10 milligram (mg) or 30 mg, or 60 mg or 120 mg.
- Part 1: GSK3389404 10 mg: Participants received a single dose of GSK3389404 10 mg by subcutaneous injection on Day 1 of Part 1.
- Part 1: GSK3389404 30 mg: Participants received a single dose of GSK3389404 30 mg by subcutaneous injection on Day 1 of Part 1.
- Part 1: GSK3389404 60 mg: Participants received a single dose of GSK3389404 60 mg by subcutaneous injection on Day 1 of Part 1.
- Part 1: GSK3389404 120 mg: Participants received a single dose of GSK3389404 120 mg by subcutaneous injection on Day 1 of Part 1.
- Part 2: Placebo: Participant received a single dose of subcutaneous injection of placebo matching with GSK3389404 30 mg or 60 mg or 120 mg once weekly (QW) for 4 weeks in Part 2.
- Part 2: GSK3389404 30 mg: Participants received a single dose of GSK3389404 30 mg by subcutaneous injection QW for 4 weeks in Part 2.
- Part 2: GSK3389404 60 mg: Participants received a single dose of GSK3389404 60 mg by subcutaneous injection QW for 4 weeks in Part 2.
- Part 2: GSK3389404 120 mg: Participants received a single dose of GSK3389404 120 mg by subcutaneous injection QW for 4 weeks in Part 2.
Period: Single-Ascending Dose(Part 1-62 Days)
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg | Part 2: Placebo | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Started | 8 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0
Completed | 8 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Multiple-Ascending Dose(Part 2-115 Days)
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg | Part 2: Placebo | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Started | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg | Part 2: Placebo | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] — Data for Part 1 is presented. Population: N=32 for Part 1
  Years
    number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 32
    (all) | 28.1 (8.22) | 27.5 (3.78) | 37.5 (12.44) | 32.8 (7.41) | 37.8 (13.41) |  |  |  |  | 32.5 (10.03)
Age, Continuous [Mean (Standard Deviation); unit: Years] — Data for Part 2 is presented. Population: N=24 for Part 2
  Years
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 24
    (all) |  |  |  |  |  | 38.0 (11.78) | 32.2 (6.91) | 40.5 (11.13) | 38.5 (12.23) | 37.3 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Male | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 6 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity, Customized: Asian-South East Asian heritage | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Race/Ethnicity, Customized: African American/African heritage | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Race/Ethnicity, Customized: White-White/Caucasian/European heritage | 8 | 3 | 4 | 6 | 6 | 4 | 5 | 3 | 6 | 45
  Race/Ethnicity, Customized: Asian-Central/South Asian heritage | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3
  Race/Ethnicity, Customized: Caribbean | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Race/Ethnicity, Customized: Caribbean British | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Non-serious Adverse Event (AE); Any Serious AE (SAE); Any AEs Leading to Discontinuation of Study Treatment (AELD) in Part 1
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention or event associated with liver injury and impaired liver function were categorized as SAE. Participants who received any of the study treatment and had any AE or SAE or AELD were considered for analysis. Safety Population comprised of all participants who received at least 1 dose of study treatment.
Time Frame: Up to 62 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Participants
  Any non-serious AE | 4 | 3 | 2 | 3 | 5
  Any SAE | 0 | 0 | 0 | 0 | 0
  AELD | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Any Non-serious AE; Any SAE; Any AELD in Part 2
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention or event associated with liver injury and impaired liver function were categorized as SAE. Participants who received any of the study treatment and had any AE or SAE or AELD were considered for analysis.
Time Frame: Up to 115 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Any non-serious AE | 3 | 5 | 2 | 4
  Any SAE | 0 | 0 | 0 | 0
  AELD | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Laboratory Values of Potential Clinical Importance in Part 1
Description: Blood samples were collected for hematology, clinical chemistry, coagulation parameters and urinalysis. Abnormalities of potential clinical importance were evaluated as per Division of Acquired Immune Deficiency Syndrome [DAIDS] table for grading the severity of adult and pediatric adverse events. Laboratory abnormalities of DAIDS Grade 1 or higher were considered as of potential clinical importance and were summarized.
Time Frame: Up to 62 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Participants | 5 | 3 | 2 | 4 | 3

4. Primary Outcome: Number of Participants With Laboratory Values of Potential Clinical Importance in Part 2
Description: Blood samples were collected for hematology, clinical chemistry, coagulation parameters and urinalysis. Abnormalities of potential clinical importance were evaluated as per DAIDS table for grading the severity of adult and pediatric adverse events. Laboratory abnormalities of DAIDS Grade 1 or higher were considered as of potential clinical importance and were summarized.
Time Frame: Up to 115 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 3 | 2 | 5 | 3

5. Primary Outcome: Change From Baseline in Complement Factor Component 3 (C3) and C4 Levels in Part 1
Description: Blood samples were collected to evaluate complement factors (C3 and C4) levels. Latest pre-dose assessment at Day 1 was considered as Baseline value. Change from Baseline was calculated as difference between minimum level (lowest of the measurements for specimens collected) observed post-dose and pre-study drug administration.
Time Frame: Day 1 (pre-dose) and up to 31 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Gram per liter (g/L)
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Gram per liter (g/L)
  C3 | -0.0811 (0.09367) | -0.0142 (0.04549) | -0.1580 (0.12739) | -0.0900 (0.07452) | -0.0412 (0.06432)
  C4 | -0.0320 (0.04107) | -0.0123 (0.01768) | -0.0600 (0.04544) | -0.0212 (0.01987) | -0.0250 (0.01979)

6. Primary Outcome: Change From Baseline in Complement Split Product C5a Levels in Part 1
Description: Blood samples were collected to evaluate complement split product C5a levels. Latest pre-dose assessment at Day 1 was considered as Baseline value. Change from Baseline was calculated as difference between maximum level (highest of the measurements for specimens collected) observed post-dose and pre-study drug administration.
Time Frame: Day 1 (pre-dose) and up to 31 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Microgram per liter (ug/L)
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Microgram per liter (ug/L) | 7.895 (4.6360) | 7.755 (8.8013) | 2.590 (1.9653) | 5.102 (18.7596) | 1.485 (2.5368)

7. Primary Outcome: Change From Baseline in Complement Split Product Bb Levels in Part 1
Description: Blood samples were collected to evaluate complement split product Bb levels. Latest pre-dose assessment at Day 1 was considered as Baseline value. Change from Baseline was calculated as difference between maximum level (highest of the measurements for specimens collected) observed post-dose and pre-study drug administration
Time Frame: Day 1 (pre-dose) and up to 31 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mg per liter (mg/L)
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
mg per liter (mg/L) | 0.8788 (1.01171) | 1.5517 (1.26063) | 0.6900 (0.48187) | 1.2900 (1.69068) | 0.3350 (0.78899)

8. Primary Outcome: Change From Baseline in Complement Factor C3 and C4 Levels in Part 2
Description: Blood samples were collected to evaluate complement factors (C3 and C4) levels. Latest pre-dose assessment at Day 1 or Day 22 was considered as Baseline value. Change from Baseline was calculated as difference between minimum level (lowest of the measurements for specimens collected each after Day 1 and Day 22 study drug administrations) observed post-dose and pre-study drug administration
Time Frame: Day 1 (pre-dose) and Day 22
Population: Safety Population
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
G/L
  C3, Day 1 | -0.0495 (0.06661) | -0.0333 (0.05961) | -0.0783 (0.04025) | -0.0293 (0.05722)
  C3, Day 22 | -0.1143 (0.07139) | -0.1013 (0.06017) | -0.0840 (0.02521) | -0.1702 (0.07908)
  C4, Day 1 | -0.0190 (0.01192) | -0.0132 (0.03511) | -0.0470 (0.02674) | -0.0135 (0.01271)
  C4, Day 22 | -0.0397 (0.02043) | -0.0405 (0.03661) | -0.0390 (0.01980) | -0.0443 (0.02805)

9. Primary Outcome: Change From Baseline in Complement Factor C5a Levels in Part 2
Description: Blood samples were collected to evaluate complement factors C5a levels. Latest pre-dose assessment at Day 1 or Day 22 was considered as Baseline value. Change from Baseline was calculated as difference between maximum level (lowest of the measurements for specimens collected each after Day 1 and Day 22 study drug administrations) observed post-dose and pre-study drug administration.
Time Frame: Day 1 (pre-dose) and Day 22
Population: Safety Population
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ug/L
  C5a, Day 1 | 3.000 (4.2895) | -1.167 (5.8963) | 2.750 (4.1563) | 11.083 (6.3907)
  C5a, Day 22 | 9.083 (4.2002) | 9.667 (10.5862) | 7.333 (2.3805) | 13.667 (9.9029)

10. Primary Outcome: Change From Baseline in Complement Factor Bb Levels in Part 2
Description: as for outcome 9
Time Frame: Day 1 (pre-dose) and Day 22
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mg/L
  Bb, Day 1 | 0.4217 (0.62669) | 0.5033 (0.76727) | 0.9700 (0.60554) | 1.2667 (0.55623)
  Bb, Day 22 | 1.4003 (0.56580) | 1.3447 (0.75517) | 0.6833 (0.57597) | 1.7340 (1.05781)

11. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at the Indicated Time Points in Part 1
Description: SBP and DBP were taken at Baseline (Day 1, pre-dose) and at 1, 2, 4, 8, 12, 24, 48 and 72 hour post dose; and on Days 8 and 30. Measurements were obtained after resting for at least 5 minutes in a semi-supine position. Baseline was defined as the last scheduled non-missing measurement taken prior to drug administration. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: Day 1 (pre-dose) and up to 30 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Millimeter of mercury (mmHg)
  DBP, 1 hour | -4.1 (6.53) | -4.4 (4.38) | -3.8 (7.36) | 1.5 (4.96) | 2.3 (4.51)
  DBP, 2 hour | -4.1 (2.46) | -3.1 (4.29) | -4.8 (3.87) | 0.6 (3.64) | -1.9 (1.86)
  DBP, 4 hour | -1.8 (3.64) | -5.6 (7.39) | -0.6 (7.39) | -0.8 (5.05) | -0.4 (5.42)
  DBP, 8 hour | -5.6 (3.66) | -5.4 (8.78) | -4.0 (7.93) | -0.7 (4.43) | -1.3 (4.34)
  DBP, 12 hour | -3.2 (7.50) | -5.8 (10.30) | -3.8 (4.01) | -1.5 (4.37) | -1.4 (4.34)
  DBP, 24 hour | -2.8 (4.29) | -4.3 (7.53) | 0.2 (9.20) | 0.1 (4.00) | -2.6 (4.11)
  DBP, 48 hour | -2.7 (4.59) | -3.3 (6.22) | -3.0 (6.87) | -1.3 (4.78) | -1.4 (2.50)
  DBP, 72 hour | -1.9 (4.38) | -2.2 (5.71) | 1.0 (7.08) | 0.5 (1.25) | -2.7 (3.19)
  DBP, Day 8 | -3.1 (5.07) | -3.4 (4.60) | -4.6 (4.53) | 0.3 (7.33) | -2.0 (2.91)
  DBP, Day 30 | -1.7 (6.28) | 0.5 (7.36) | -5.1 (6.92) | 2.1 (7.26) | -0.3 (4.32)
  SBP, 1 hour | -2.0 (7.65) | -4.0 (3.85) | -0.8 (8.55) | 1.8 (6.22) | 0.2 (6.18)
  SBP, 2 hour | -0.7 (5.63) | 0.3 (5.89) | 2.2 (8.08) | 2.1 (5.51) | 4.9 (3.67)
  SBP, 4 hour | -1.5 (4.58) | -5.5 (6.42) | -0.9 (4.32) | -4.6 (7.68) | 0.3 (5.94)
  SBP, 8 hour | -1.6 (6.27) | -4.6 (11.61) | -2.3 (5.31) | 1.2 (5.61) | 4.1 (4.19)
  SBP, 12 hour | 1.6 (10.73) | -5.5 (10.15) | 0.8 (4.58) | -1.5 (7.04) | 2.2 (3.54)
  SBP, 24 hour | -4.0 (6.40) | -4.8 (6.42) | 3.1 (8.30) | -0.6 (6.39) | -0.9 (2.69)
  SBP, 48 hour | -0.4 (6.84) | -6.8 (5.48) | -5.0 (3.89) | -1.7 (4.07) | -2.1 (4.03)
  SBP, 72 hour | -1.4 (5.08) | -2.8 (8.29) | 4.6 (9.89) | 0.6 (4.24) | -1.5 (2.95)
  SBP, Day 8 | -0.3 (7.41) | -4.8 (4.87) | -2.7 (5.98) | 0.5 (6.61) | 0.5 (3.48)
  SBP, Day 30 | 2.7 (8.17) | -1.7 (8.21) | -0.1 (6.84) | -0.9 (4.75) | 5.9 (3.50)

12. Primary Outcome: Change From Baseline in Pulse Rate (PR) at the Indicated Time Points in Part 1
Description: Pulse rate was taken at Baseline (Day 1, pre-dose) and at 1, 2, 4, 8, 12, 24, 48 and 72 hour post dose; and on Days 8 and 30. Measurements were obtained after resting for at least 5 minutes in a semi-supine position. Baseline was defined as the last scheduled non-missing measurement taken prior to drug administration. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: Day 1 (pre-dose) and up to 30 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Beats per minute (bpm)
  PR, 1 hour | 0.2 (3.20) | 0.3 (5.49) | -2.0 (3.19) | 1.5 (5.43) | -3.2 (6.63)
  PR, 2 hour | 1.6 (3.68) | 4.0 (12.68) | 2.3 (4.54) | 3.8 (6.00) | -2.3 (8.82)
  PR, 4 hour | 0.4 (5.83) | -0.5 (7.68) | -1.9 (3.24) | 0.2 (5.53) | 0.7 (9.37)
  PR, 8 hour | 1.5 (4.46) | 1.2 (4.50) | 1.9 (2.63) | 4.8 (5.89) | 1.3 (6.76)
  PR, 12 hour | 6.9 (12.49) | 1.6 (5.04) | 2.3 (4.19) | 8.6 (8.12) | -0.7 (8.35)
  PR, 24 hour | -1.9 (4.49) | -1.6 (9.89) | 1.4 (7.17) | -1.3 (5.49) | -0.9 (10.07)
  PR, 48 hour | 1.8 (10.74) | 0.2 (9.79) | 1.4 (4.46) | 2.3 (5.10) | -0.6 (6.61)
  PR, 72 hour | 3.7 (4.85) | 1.0 (5.26) | 4.0 (3.47) | 5.3 (5.39) | 0.3 (9.90)
  PR, Day 8 | 3.5 (5.55) | 0.4 (6.34) | 1.4 (2.58) | 6.0 (7.36) | 1.5 (9.03)
  PR, Day 30 | 2.0 (6.53) | 4.3 (11.94) | 0.2 (5.36) | 6.3 (6.19) | -1.1 (9.67)

13. Primary Outcome: Change From Baseline in Respiratory Rate (RR) at the Indicated Time Points in Part 1
Description: Respiratory rate was taken at Baseline (Day 1, pre-dose) and at 1, 2, 4, 8, 12, 24, 48 and 72 hour post dose; and on Days 8 and 30. Baseline was defined as the last scheduled non-missing measurement taken prior to drug administration. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: Day 1 (pre-dose) and up to 30 days
Population: Safety Population. Only data available at the specified time points was analyzed. (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Breaths per minute
  RR, 1 hour, n=8, 6, 6, 6, 6 | -0.5 (2.14) | -1.3 (1.86) | 0.8 (3.54) | 1.5 (2.59) | 0.7 (3.67)
  RR, 2 hour, n=8, 6, 6, 6, 6 | -0.3 (2.38) | 0.3 (3.14) | -2.7 (2.66) | 1.0 (4.15) | -1.7 (1.63)
  RR, 4 hour, n=8, 6, 6, 5, 6: number analyzed (Participants) | 8 | 6 | 6 | 5 | 6
  RR, 4 hour, n=8, 6, 6, 5, 6 | -0.8 (3.01) | -0.2 (2.14) | 0.0 (2.90) | 0.4 (5.50) | 0.2 (3.31)
  RR, 8 hour, n=8, 6, 6, 6, 6 | -0.1 (2.95) | -0.5 (1.87) | -1.0 (3.79) | -1.2 (3.87) | -2.2 (1.83)
  RR, 12 hour, n=8, 6, 6, 6, 6 | -0.3 (2.19) | 0.8 (1.60) | -0.5 (2.59) | 0.0 (3.10) | 0.0 (1.41)
  RR, 24 hour, n=8, 6, 6, 6, 6 | -0.6 (2.62) | -0.3 (2.94) | -2.2 (3.54) | 0.5 (1.52) | -0.7 (1.75)
  RR, 48 hour, n=8, 6, 6, 6, 6 | -0.5 (3.12) | -0.8 (2.32) | -2.0 (3.74) | 3.0 (3.29) | 1.7 (1.63)
  RR, 72 hour, n=8, 6, 6, 6, 6 | -0.5 (3.07) | 0.7 (3.44) | 0.0 (3.52) | 0.8 (3.66) | -1.7 (2.25)
  RR, Day 8, n=8, 6, 6, 6, 6 | -0.6 (3.20) | -1.3 (1.51) | -1.5 (4.72) | 1.0 (2.97) | -1.0 (2.68)
  RR, Day 30, n=8, 6, 6, 6, 6 | 1.0 (1.69) | 0.0 (1.41) | -0.7 (3.44) | -0.7 (3.50) | -0.3 (2.25)

14. Primary Outcome: Change From Baseline in Body Temperature at the Indicated Time Points in Part 1
Description: Temperature was taken at Baseline (Day 1, pre-dose) and at 1, 2, 4, 8, 12, 24, 48 and 72 hour post dose; and on Days 8 and 30. Baseline was defined as the last scheduled non-missing measurement taken prior to drug administration. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: Day 1 (pre-dose) and up to 30 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Degree Celsius
  Temperature, 1 hour | 0.06 (0.185) | 0.00 (0.237) | 0.05 (0.122) | 0.10 (0.276) | 0.10 (0.200)
  Temperature, 2 hour | 0.04 (0.288) | -0.02 (0.147) | 0.02 (0.172) | -0.15 (0.243) | 0.05 (0.243)
  Temperature, 4 hour | 0.14 (0.213) | 0.08 (0.319) | 0.05 (0.217) | -0.02 (0.264) | 0.08 (0.194)
  Temperature, 8 hour | 0.24 (0.297) | -0.02 (0.279) | 0.20 (0.126) | 0.18 (0.147) | 0.23 (0.288)
  Temperature, 12 hour | 0.18 (0.255) | 0.03 (0.234) | -0.03 (0.137) | 0.12 (0.204) | 0.08 (0.232)
  Temperature, 24 hour | -0.01 (0.290) | -0.10 (0.167) | -0.05 (0.152) | 0.07 (0.197) | -0.03 (0.350)
  Temperature, 48 hour | 0.00 (0.434) | -0.10 (0.210) | 0.03 (0.121) | 0.02 (0.248) | -0.10 (0.276)
  Temperature, 72 hour | 0.06 (0.220) | -0.07 (0.250) | 0.07 (0.225) | 0.07 (0.175) | -0.03 (0.197)
  Temperature, Day 8 | 0.00 (0.233) | -0.08 (0.319) | 0.00 (0.200) | -0.20 (0.228) | 0.05 (0.138)
  Temperature, Day 30 | -0.04 (0.177) | -0.07 (0.216) | 0.00 (0.190) | -0.07 (0.225) | -0.12 (0.436)

15. Primary Outcome: Change From Baseline in SBP and DBP at the Indicated Time Points in Part 2
Description: SBP and DBP were taken at Baseline (Day 1, pre-dose) and at 1, 2, 4, 6, 8, 12, 24, 48 and 72 hour post Day 1 dose; on Days 8 and 15; Day 22 (pre-dose) and at 1, 4, 6, 12, 24, 48 and 72 hours post Day 22 dose; on Days 29, 36, 50, 71 and at Follow-up visit (Day 113 +- 2 days). Measurements were obtained after resting for at least 5 minutes in a semi-supine position. Baseline was defined as the last scheduled non-missing measurement taken prior to drug administration. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: Day 1 (pre-dose) and up to 115 days
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mmHg
  DBP, Day 1, 1 hour, n=6, 6, 6, 6 | 0.5 (4.75) | 5.7 (4.83) | -1.8 (3.49) | -2.4 (4.26)
  DBP, Day 1, 2 hour, n=6, 6, 6, 6 | 2.1 (5.56) | -0.1 (4.83) | -0.8 (6.74) | -1.6 (3.47)
  DBP, Day 1, 4 hour, n=6, 6, 6, 6 | -2.1 (5.54) | -5.1 (6.25) | -4.6 (5.86) | -8.0 (3.69)
  DBP, Day 1, 6 hour, n=6, 6, 6, 6 | -5.3 (5.51) | -2.6 (6.90) | -3.5 (5.03) | -5.1 (3.37)
  DBP, Day 1, 8 hour, n=6, 6, 6, 6 | -0.2 (6.66) | 1.4 (4.12) | -3.0 (8.63) | -4.1 (3.51)
  DBP, Day 1, 12 hour, n=6, 6, 6, 6 | -4.4 (7.17) | -2.6 (4.49) | -7.7 (5.97) | -4.4 (4.75)
  DBP, Day 2, 24 hour, n=6, 6, 6, 6 | 2.6 (6.29) | 0.9 (3.36) | -3.0 (4.87) | -2.1 (2.10)
  DBP, Day 3, 48 hour, n=6, 6, 6, 6 | -0.2 (5.41) | 2.6 (5.55) | -4.8 (5.24) | -2.6 (4.76)
  DBP, Day 4, 72 hour, n=6, 6, 6, 6 | 1.6 (5.77) | -6.1 (6.56) | -1.9 (3.09) | -0.1 (4.13)
  DBP, Day 8, n=6, 6, 6, 6 | 1.6 (7.61) | 1.9 (5.59) | -2.6 (3.82) | -3.0 (5.66)
  DBP, Day 15, n=6, 6, 6, 6 | 2.9 (11.22) | 5.5 (3.60) | 2.6 (6.70) | -3.1 (3.82)
  DBP, Day 22, pre-dose, n=6, 6, 6, 6 | 1.0 (7.07) | -3.8 (4.91) | -3.1 (1.66) | -2.2 (2.37)
  DBP, Day 22, 1 hour, n=6, 6, 6, 6 | 2.6 (6.79) | -0.8 (7.56) | -2.3 (6.39) | -1.8 (3.44)
  DBP, Day 22, 4 hour, n=6, 6, 6, 6 | -4.0 (7.53) | -0.3 (6.34) | -4.8 (6.46) | -3.4 (4.48)
  DBP, Day 22, 6 hour, n=6, 6, 6, 6 | -4.5 (6.22) | 0.1 (5.44) | -9.3 (8.96) | -4.2 (6.42)
  DBP, Day 22, 8 hour, n=6, 6, 6, 6 | -0.3 (5.82) | -2.8 (6.29) | -4.4 (7.14) | -1.2 (2.55)
  DBP, Day 22, 12 hour, n=6, 6, 6, 6 | -0.1 (7.80) | -2.9 (3.01) | -7.0 (9.15) | -2.6 (4.15)
  DBP, Day 23, 24 hour, n=6, 6, 6, 6 | 0.7 (8.59) | -4.2 (6.14) | -4.5 (4.00) | -0.6 (4.08)
  DBP, Day 24, 48 hour, n=6, 6, 6, 6 | -0.6 (5.84) | -2.8 (5.32) | -1.7 (4.30) | -0.9 (8.38)
  DBP, Day 25, 72 hour, n=6, 6, 6, 6 | 1.3 (6.71) | 0.7 (3.88) | 0.4 (2.83) | 0.1 (5.00)
  DBP, Day 29, n=6, 6, 6, 6 | 0.6 (9.06) | 5.7 (7.45) | 1.1 (4.70) | -2.9 (4.30)
  DBP, Day 36, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  DBP, Day 36, n=6, 6, 6, 5 | -0.8 (8.10) | 4.3 (7.05) | 1.7 (4.67) | 2.6 (5.09)
  DBP, Day 50, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  DBP, Day 50, n=6, 6, 6, 5 | 5.8 (3.93) | 9.7 (7.90) | 2.9 (4.39) | -0.1 (6.22)
  DBP, Day 71, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  DBP, Day 71, n=6, 6, 6, 5 | 3.2 (6.27) | 8.9 (6.31) | 2.4 (3.94) | 4.0 (2.22)
  DBP, Follow-up, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  DBP, Follow-up, n=6, 6, 6, 5 | 3.7 (6.38) | 2.2 (6.54) | 4.3 (3.85) | 7.7 (1.75)
  SBP, Day 1, 1 hour, n=6, 6, 6, 6 | 1.2 (5.55) | 3.4 (6.83) | 1.1 (5.35) | 5.3 (4.17)
  SBP, Day 1, 2 hour, n=6, 6, 6, 6 | 0.7 (5.95) | 0.5 (2.99) | -0.6 (3.38) | 3.9 (8.89)
  SBP, Day 1, 4 hour, n=6, 6, 6, 6 | -2.6 (6.36) | -2.6 (2.16) | -4.6 (6.57) | 0.4 (4.28)
  SBP, Day 1, 6 hour, n=6, 6, 6, 6 | -3.6 (6.23) | -0.9 (3.71) | -1.6 (6.54) | 5.4 (6.67)
  SBP, Day 1, 8 hour, n=6, 6, 6, 6 | 0.3 (3.26) | 0.6 (3.65) | 0.4 (10.56) | 5.8 (6.37)
  SBP, Day 1, 12 hour, n=6, 6, 6, 6 | -0.1 (6.39) | -0.4 (5.32) | -2.9 (7.54) | 5.8 (4.11)
  SBP, Day 2, 24 hour, n=6, 6, 6, 6 | 3.0 (6.25) | -0.1 (4.35) | 0.4 (4.95) | 2.4 (2.83)
  SBP, Day 3, 48 hour, n=6, 6, 6, 6 | 0.7 (8.69) | 1.5 (6.13) | -2.4 (6.34) | 5.0 (4.38)
  SBP, Day 4, 72 hour, n=6, 6, 6, 6 | 3.9 (4.96) | -3.7 (6.64) | 0.2 (7.29) | 7.5 (3.32)
  SBP, Day 8, n=6, 6, 6, 6 | -0.7 (7.45) | -1.7 (6.25) | -4.4 (5.97) | 2.8 (7.24)
  SBP, Day 15, n=6, 6, 6, 6 | 3.5 (10.88) | 4.6 (7.93) | -2.3 (6.47) | 1.5 (5.47)
  SBP, Day 22, pre-dose, n=6, 6, 6, 6 | -1.1 (9.18) | -4.6 (5.69) | -4.0 (2.60) | -1.1 (5.65)
  SBP, Day 22, 1 hour, n=6, 6, 6, 6 | 1.7 (6.34) | -4.6 (4.41) | -1.6 (2.20) | 3.2 (7.34)
  SBP, Day 22, 4 hour, n=6, 6, 6, 6 | -0.3 (6.11) | -2.0 (4.70) | -4.2 (5.24) | 2.5 (4.99)
  SBP, Day 22, 6 hour, n=6, 6, 6, 6 | -2.4 (7.57) | -2.7 (2.55) | -6.1 (7.77) | 1.3 (5.49)
  SBP, Day 22, 8 hour, n=6, 6, 6, 6 | -0.3 (5.73) | -5.9 (2.98) | -5.4 (6.27) | 0.6 (4.57)
  SBP, Day 22, 12 hour, n=6, 6, 6, 6 | 4.9 (6.14) | 0.1 (3.22) | -5.2 (8.57) | 5.2 (4.07)
  SBP, Day 23, 24 hour, n=6, 6, 6, 6 | 0.8 (8.50) | -5.7 (3.77) | -1.2 (5.67) | 4.9 (6.35)
  SBP, Day 24, 48 hour, n=6, 6, 6, 6 | 0.3 (3.79) | -7.4 (4.48) | -0.8 (5.02) | 2.8 (5.29)
  SBP, Day 25, 72 hour, n=6, 6, 6, 6 | 1.2 (5.37) | -1.0 (3.48) | 4.4 (5.69) | 5.0 (3.87)
  SBP, Day 29, n=6, 6, 6, 6 | 0.3 (6.24) | 6.8 (7.69) | -1.0 (4.68) | 1.9 (5.57)
  SBP, Day 36, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  SBP, Day 36, n=6, 6, 6, 5 | -2.8 (9.99) | 4.2 (7.35) | 0.7 (6.11) | 3.2 (3.89)
  SBP, Day 50, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  SBP, Day 50, n=6, 6, 6, 5 | 8.1 (6.28) | 3.9 (4.47) | -0.7 (7.20) | 2.5 (2.32)
  SBP, Day 71, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  SBP, Day 71, n=6, 6, 6, 5 | 1.1 (7.49) | 4.9 (7.81) | 4.1 (7.42) | 7.4 (5.34)
  SBP, Follow-up, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  SBP, Follow-up, n=6, 6, 6, 5 | 4.8 (8.05) | -2.1 (7.16) | 10.0 (5.98) | 11.5 (5.29)

16. Primary Outcome: Change From Baseline in PR at the Indicated Time Points in Part 2
Description: Pulse rate was taken at Baseline (Day 1, pre-dose) and at 1, 2, 4, 6, 8, 12, 24, 48 and 72 hour post Day 1 dose; on Days 8 and 15; Day 22 (pre-dose) and at 1, 4, 6, 12, 24, 48 and 72 hours post Day 22 dose; on Days 29, 36, 50, 71 and at Follow-up visit (Day 113+- 2 days). Measurements were obtained after resting for at least 5 minutes in a semi-supine position. Baseline was defined as the last scheduled non-missing measurement taken prior to drug administration. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: Day 1 (pre-dose) and up to 115 days
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
bpm
  PR, Day 1, 1 hour, n=6, 6, 6, 6 | -1.5 (7.15) | 0.5 (3.80) | 0.3 (1.54) | -2.4 (2.09)
  PR, Day 1, 2 hour, n=6, 6, 6, 6 | 0.4 (4.57) | -1.6 (6.79) | 2.9 (4.17) | -1.1 (3.81)
  PR, Day 1, 4 hour, n=6, 6, 6, 6 | 4.7 (4.13) | 4.6 (5.99) | 6.6 (3.75) | 2.4 (2.79)
  PR, Day 1, 6 hour, n=6, 6, 6, 6 | 6.4 (2.38) | 5.8 (7.12) | 7.9 (3.27) | 6.6 (3.93)
  PR, Day 1, 8 hour, n=6, 6, 6, 6 | 0.4 (1.83) | 3.5 (5.39) | 7.8 (6.99) | 0.5 (3.91)
  PR, Day 1, 12 hour, n=6, 6, 6, 6 | 4.0 (3.29) | 7.2 (7.13) | 7.8 (6.09) | 3.9 (4.59)
  PR, Day 2, 24 hour, n=6, 6, 6, 6 | 0.6 (4.62) | -2.4 (4.84) | 2.4 (3.33) | -1.1 (2.39)
  PR, Day 3, 48 hour, n=6, 6, 6, 6 | 3.8 (4.90) | 4.3 (9.58) | 6.2 (5.70) | -0.1 (2.93)
  PR, Day 4, 72 hour, n=6, 6, 6, 6 | 10.1 (8.83) | 5.7 (5.30) | 10.8 (8.06) | 4.0 (7.05)
  PR, Day 8, n=6, 6, 6, 6 | 0.5 (3.11) | 1.6 (8.20) | 7.1 (6.86) | -1.6 (2.55)
  PR, Day 15, n=6, 6, 6, 6 | -0.2 (10.22) | 4.9 (12.25) | 2.4 (3.52) | -5.7 (6.04)
  PR, Day 22, pre-dose, n=6, 6, 6, 6 | 2.7 (6.80) | 8.0 (14.84) | 1.5 (1.59) | -2.9 (4.51)
  PR, Day 22, 1 hour, n=6, 6, 6, 6 | 1.4 (4.84) | -3.1 (4.22) | 2.2 (3.35) | -3.2 (7.19)
  PR, Day 22, 4 hour, n=6, 6, 6, 6 | 6.0 (4.01) | 4.3 (5.87) | 11.5 (10.74) | 2.6 (6.63)
  PR, Day 22, 6 hour, n=6, 6, 6, 6 | 7.2 (3.75) | 3.8 (1.81) | 8.6 (3.98) | 2.4 (5.99)
  PR, Day 22, 8 hour, n=6, 6, 6, 6 | 2.2 (6.26) | -1.6 (5.59) | 5.7 (3.61) | -2.1 (5.06)
  PR, Day 22, 12 hour, n=6, 6, 6, 6 | 6.4 (4.03) | 5.4 (4.64) | 9.3 (4.47) | 7.9 (7.02)
  PR, Day 23, 24 hour, n=6, 6, 6, 6 | 3.6 (3.46) | 0.0 (4.92) | 4.6 (6.63) | 0.7 (7.64)
  PR, Day 24, 48 hour, n=6, 6, 6, 6 | 4.1 (2.88) | -1.0 (4.85) | 3.6 (3.79) | 2.9 (9.40)
  PR, Day 25, 72 hour, n=6, 6, 6, 6 | 8.7 (10.05) | 7.1 (5.05) | 7.0 (4.94) | 4.3 (7.77)
  PR, Day 29, n=6, 6, 6, 6 | 8.4 (4.76) | 6.9 (8.33) | 5.0 (1.14) | -0.6 (7.41)
  PR, Day 36, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  PR, Day 36, n=6, 6, 6, 5 | 4.1 (6.54) | 5.4 (7.51) | 3.8 (6.10) | -3.2 (13.57)
  PR, Day 50, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  PR, Day 50, n=6, 6, 6, 5 | 9.9 (4.85) | 1.1 (2.09) | 2.2 (6.51) | -7.0 (6.34)
  PR, Day 71, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  PR, Day 71, n=6, 6, 6, 5 | 6.1 (2.74) | 5.1 (7.39) | 6.0 (2.04) | -1.9 (6.93)
  PR, Follow-up, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  PR, Follow-up, n=6, 6, 6, 5 | 6.1 (6.79) | 2.7 (5.08) | 6.0 (4.23) | 2.0 (5.71)

17. Primary Outcome: Change From Baseline in RR at the Indicated Time Points in Part 2
Description: Respiratory rate was taken at Baseline (Day 1, pre-dose) and at 1, 2, 4, 6, 8, 12, 24, 48 and 72 hour post Day 1 dose; on Days 8 and 15; Day 22 (pre-dose) and at 1, 4, 6, 12, 24, 48 and 72 hours post Day 22 dose; on Days 29, 36, 50, 71 and at Follow-up visit (Day 113+- 2 days). Baseline was defined as the last scheduled non-missing measurement taken prior to drug administration. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: Day 1 (pre-dose) and up to 115 days
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Breaths per minute
  RR, Day 1, 1 hour, n=6, 6, 6, 6 | -0.3 (1.97) | 0.7 (2.73) | 0.0 (1.26) | 0.5 (1.97)
  RR, Day 1, 2 hour, n=6, 6, 6, 6 | -0.3 (1.97) | -0.3 (2.34) | 0.7 (1.63) | 0.5 (1.22)
  RR, Day 1, 4 hour, n=6, 6, 6, 6 | 0.0 (3.35) | 1.0 (3.52) | -0.7 (2.42) | -0.5 (0.84)
  RR, Day 1, 6 hour, n=6, 6, 6, 6 | -0.3 (2.66) | 1.3 (4.13) | 2.0 (2.53) | -0.5 (0.84)
  RR, Day 1, 8 hour, n=6, 6, 6, 6 | -0.7 (2.73) | 1.3 (3.01) | 0.7 (2.42) | 0.8 (1.83)
  RR, Day 1, 12 hour, n=6, 6, 6, 6 | 2.0 (3.79) | 1.7 (2.66) | 3.3 (2.42) | 0.5 (2.95)
  RR, Day 2, 24 hour, n=6, 6, 6, 6 | 0.7 (2.42) | 1.0 (2.10) | -1.7 (1.51) | -0.5 (0.84)
  RR, Day 3, 48 hour, n=6, 6, 6, 6 | -1.0 (2.10) | -0.3 (2.34) | -1.0 (2.76) | -0.8 (1.60)
  RR, Day 4, 72 hour, n=6, 6, 6, 6 | 0.8 (2.71) | 1.3 (3.67) | 0.3 (3.44) | -0.2 (1.33)
  RR, Day 8, n=6, 6, 6, 6 | 1.3 (1.63) | -0.3 (3.88) | 1.3 (3.72) | -0.8 (3.13)
  RR, Day 15, n=6, 6, 6, 6 | 0.7 (1.63) | 1.5 (1.76) | 0.7 (2.42) | -0.8 (3.13)
  RR, Day 22, pre-dose, n=6, 6, 6, 6 | 0.0 (1.79) | 0.7 (2.42) | -1.0 (2.45) | -0.5 (1.97)
  RR, Day 22, 1 hour, n=6, 6, 6, 6 | 0.7 (3.27) | 0.3 (3.88) | -0.3 (3.88) | 0.5 (1.52)
  RR, Day 22, 4 hour, n=6, 6, 6, 6 | -0.7 (1.63) | 1.8 (4.02) | -1.0 (3.74) | 0.8 (0.98)
  RR, Day 22, 6 hour, n=6, 6, 6, 6 | 1.0 (2.10) | 2.3 (3.88) | 3.0 (2.76) | 0.2 (2.56)
  RR, Day 22, 8 hour, n=6, 6, 6, 6 | 1.7 (1.97) | 2.7 (3.50) | -0.7 (2.07) | -0.8 (1.83)
  RR, Day 22, 12 hour, n=6, 6, 6, 6 | 2.3 (3.20) | 4.3 (3.20) | 1.0 (2.10) | -1.5 (2.35)
  RR, Day 23, 24 hour, n=6, 6, 6, 6 | 0.7 (3.50) | 1.3 (2.73) | -0.3 (2.94) | -0.5 (0.84)
  RR, Day 24, 48 hour, n=6, 6, 6, 6 | 1.0 (3.03) | 1.7 (2.94) | -0.3 (2.66) | -0.5 (2.66)
  RR, Day 25, 72 hour, n=6, 6, 6, 6 | 1.0 (2.76) | 2.7 (2.42) | -0.7 (3.01) | -1.5 (1.22)
  RR, Day 29, n=6, 6, 6, 6 | 0.7 (1.63) | 1.3 (2.73) | -1.0 (1.67) | -0.2 (1.33)
  RR, Day 36, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  RR, Day 36, n=6, 6, 6, 5 | 0.0 (3.10) | 0.7 (3.27) | 0.0 (3.35) | -1.0 (1.73)
  RR, Day 50, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  RR, Day 50, n=6, 6, 6, 5 | 0.5 (3.56) | 1.0 (3.74) | -0.7 (3.27) | -0.2 (1.48)
  RR, Day 71, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  RR, Day 71, n=6, 6, 6, 5 | 0.2 (2.40) | 1.3 (1.03) | 0.0 (4.00) | 0.6 (1.34)
  RR, Follow-up, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  RR, Follow-up, n=6, 6, 6, 5 | -1.7 (1.51) | -1.0 (1.67) | -0.7 (3.50) | 0.6 (2.61)

18. Primary Outcome: Change From Baseline in Body Temperature at the Indicated Time Points in Part 2
Description: Body temperature was taken at Baseline (Day 1, pre-dose) and at 1, 2, 4, 6, 8, 12, 24, 48 and 72 hour post Day 1 dose; on Days 8 and 15; Day 22 (pre-dose) and at 1, 4, 6, 12, 24, 48 and 72 hours post Day 22 dose; on Days 29, 36, 50, 71 and at Follow-up visit (Day 113+- 2 days). Baseline was defined as the last scheduled non-missing measurement taken prior to drug administration. Change from Baseline was calculated as value at indicated time point minus Baseline value.
Time Frame: Day 1 (pre-dose) and up to 115 days
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Part 2: Placebo | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Degree Celsius
  Temperature, Day 1, 1 hour, n=6, 6, 6, 6 | 0.27 (0.388) | 0.15 (0.288) | -0.05 (0.176) | 0.02 (0.440)
  Temperature, Day 1, 2 hour, n=6, 6, 6, 6 | 0.20 (0.167) | -0.02 (0.256) | 0.05 (0.187) | -0.02 (0.240)
  Temperature, Day 1, 4 hour, n=6, 6, 6, 6 | 0.40 (0.110) | 0.35 (0.308) | 0.02 (0.117) | 0.15 (0.432)
  Temperature, Day 1, 6 hour, n=6, 6, 6, 6 | 0.28 (0.325) | 0.38 (0.454) | 0.10 (0.237) | 0.20 (0.358)
  Temperature, Day 1, 8 hour, n=6, 6, 6, 6 | 0.20 (0.228) | 0.43 (0.408) | -0.13 (0.320) | 0.33 (0.557)
  Temperature, Day 1, 12 hour, n=6, 6, 6, 6 | 0.22 (0.147) | 0.50 (0.369) | -0.15 (0.295) | 0.20 (0.390)
  Temperature, Day 2, 24 hour, n=6, 6, 6, 6 | 0.05 (0.321) | -0.10 (0.379) | -0.18 (0.223) | -0.15 (0.138)
  Temperature, Day 3, 48 hour, n=6, 6, 6, 6 | 0.05 (0.442) | 0.15 (0.489) | -0.22 (0.204) | -0.32 (0.313)
  Temperature, Day 4, 72 hour, n=6, 6, 6, 6 | -0.05 (0.362) | 0.28 (0.595) | 0.30 (0.210) | -0.02 (0.417)
  Temperature, Day 8, n=6, 6, 6, 6 | 0.02 (0.436) | 0.05 (0.235) | 0.10 (0.283) | -0.20 (0.424)
  Temperature, Day 15, n=6, 6, 6, 6 | -0.23 (0.446) | 0.08 (0.376) | -0.05 (0.197) | -0.12 (0.366)
  Temperature, Day 22, pre-dose, n=6, 6, 6, 6 | 0.08 (0.488) | -0.02 (0.331) | -0.22 (0.183) | -0.23 (0.082)
  Temperature, Day 22, 1 hour, n=6, 6, 6, 6 | 0.15 (0.266) | -0.15 (0.315) | -0.07 (0.175) | -0.20 (0.303)
  Temperature, Day 22, 4 hour, n=6, 6, 6, 6 | 0.38 (0.422) | 0.13 (0.513) | 0.07 (0.242) | -0.18 (0.366)
  Temperature, Day 22, 6 hour, n=6, 6, 6, 6 | 0.22 (0.306) | 0.28 (0.248) | 0.17 (0.163) | -0.02 (0.293)
  Temperature, Day 22, 8 hour, n=6, 6, 6, 6 | 0.25 (0.217) | 0.23 (0.367) | -0.05 (0.243) | -0.02 (0.214)
  Temperature, Day 22, 12 hour, n=6, 6, 6, 6 | 0.22 (0.366) | 0.08 (0.299) | 0.27 (0.344) | 0.22 (0.147)
  Temperature, Day 23, 24 hour, n=6, 6, 6, 6 | 0.18 (0.366) | 0.15 (0.536) | -0.13 (0.216) | -0.12 (0.279)
  Temperature, Day 24, 48 hour, n=6, 6, 6, 6 | 0.12 (0.417) | 0.00 (0.352) | -0.08 (0.098) | -0.13 (0.432)
  Temperature, Day 25, 72 hour, n=6, 6, 6, 6 | 0.10 (0.276) | 0.20 (0.562) | 0.12 (0.445) | -0.20 (0.276)
  Temperature, Day 29, n=6, 6, 6, 6 | -0.38 (0.366) | -0.05 (0.187) | -0.15 (0.266) | -0.23 (0.250)
  Temperature, Day 36, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  Temperature, Day 36, n=6, 6, 6, 5 | 0.22 (0.271) | 0.03 (0.350) | -0.20 (0.385) | -0.16 (0.378)
  Temperature, Day 50, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  Temperature, Day 50, n=6, 6, 6, 5 | 0.02 (0.325) | -0.07 (0.480) | -0.37 (0.121) | 0.04 (0.416)
  Temperature, Day 71, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  Temperature, Day 71, n=6, 6, 6, 5 | -0.18 (0.286) | -0.13 (0.378) | -0.53 (0.280) | -0.34 (0.305)
  Temperature, Follow-up, n=6, 6, 6, 5: number analyzed (Participants) | 6 | 6 | 6 | 5
  Temperature, Follow-up, n=6, 6, 6, 5 | -0.18 (0.479) | 0.08 (0.397) | -0.12 (0.293) | -0.02 (0.259)

19. Primary Outcome: Number of Participants With 12-lead Electrocardiogram (ECG) Findings in Part 1
Description: 12-lead ECGs were recorded at Baseline (Day 1, pre-dose) and at 1, 4, 8, 12, 24 and 48 hour post dose; and on Days 8 and 30. Measurements were obtained after resting for at least 5 minutes in a supine position. Baseline was defined as the last scheduled non-missing measurement taken prior to drug administration. Change from Baseline was calculated as value at indicated time point minus Baseline value. Number of participants with worst change from Baseline in ECG have been presented as clinically significant (CS) change or not a clinically significant (NCS) change.
Time Frame: Day 1 (pre-dose) and up to 31 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
Participants
  CS | 0 | 0 | 0 | 0 | 0
  NCS | 2 | 0 | 1 | 1 | 3

20. Primary Outcome: Area Under the Plasma Concentration Curve (AUC) From Time Zero to Infinity [AUC (0-inf)], AUC From Time Zero to the Time of Last Quantifiable Concentration [AUC(0-t)], AUC From Time Zero to 24 Hours [AUC(0-24)] of GSK3389404 After Single Dose in Part 1
Description: Blood samples were collected to evaluate AUC (0-inf), AUC (0-t) and AUC (0-24) of GSK3389404 on Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 30 post-dose. Pharmacokinetic Concentration Population was defined as participants who underwent plasma PK sampling and had evaluable PK assay results post-dose.
Time Frame: Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 30 post-dose
Population: Pharmacokinetic Concentration Population
Measure: Mean (Standard Deviation); unit: Nanogram*hour per milliliter(ng*hour/mL)
Arm/Group | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6
Nanogram*hour per milliliter(ng*hour/mL)
  AUC (0-inf) | 632 (171.59) | 2080 (801.85) | 4750 (1450.8) | 8150 (3204.5)
  AUC (0-t) | 484 (80.962) | 1770 (961.03) | 3710 (1485.6) | 7440 (2844.8)
  AUC (0-24) | 592 (105.91) | 1970 (855.08) | 4330 (1313.5) | 7950 (3264.9)

21. Primary Outcome: Maximum Observed Concentration (Cmax), Observed Concentration at 24 Hours (C24) and at 168 Hours (C168) of GSK3389404 Following Single Dose in Part 1
Description: Blood samples were collected to evaluate Cmax, C24 and C168 of GSK3389404 on Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 30 post-dose.
Time Frame: Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 30 post-dose
Population: Pharmacokinetic Concentration Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6
ng/mL
  Cmax | 92.5 (23.622) | 350 (257.48) | 584 (366.96) | 889 (496.73)
  C24 | 0.00 (0.0000) | 0.00 (0.0000) | 3.33 (8.1650) | 18.7 (17.781)
  C168 | 0.00 (0.0000) | 0.00 (0.0000) | 0.00 (0.0000) | 0.00 (0.0000)

22. Primary Outcome: Time to Maximum Observed Concentration (Tmax), Terminal Half-life (T1/2) and Lag Time (Tlag) of GSK3389404 Following Single Dose in Part 1
Description: Blood samples were collected to evaluate Tmax, T1/2 and Tlag of GSK3389404 on Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 30 post-dose.
Time Frame: Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 30 post-dose
Population: Pharmacokinetic Concentration Population
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6
Hour
  Tmax | 1.60 (1.20) | 1.74 (0.48) | 2.67 (1.37) | 3.83 (0.41)
  T1/2 | 4.55 (3.3937) | 4.67 (3.5530) | 6.07 (3.9531) | 4.27 (1.2281)
  Tlag | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

23. Primary Outcome: Apparent SC Plasma Clearance (CL/F) of GSK3389404 Following Single Dose in Part 1
Description: Blood samples were collected to evaluate CL/F of GSK3389404 on Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 30 post-dose.
Time Frame: Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 30 post-dose
Population: Pharmacokinetic Concentration Population
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6
Liter per hour | 16.8 (4.2805) | 15.8 (4.6710) | 13.6 (3.6934) | 16.2 (4.7050)

24. Primary Outcome: AUC (0-t), AUC(0-24), AUC From Time Zero to 168 Hours Post-dose [AUC(0-168)] and AUC (0-inf) of GSK3389404 Following Single Dose on Day 1 of Part 2
Description: Blood samples were collected to evaluate AUC (0-t), AUC (0-24), AUC (0-168) and AUC (0-inf) of GSK3389404 on Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 15 post-dose.
Time Frame: Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 15 post-dose
Population: Pharmacokinetic Concentration Population. Only data available at the specified time points was analyzed. (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6
ng*hour/mL
  AUC (0-t), n=6, 6, 6 | 1300 (286.51) | 4150 (1103.1) | 7970 (3082.7)
  AUC (0-24), n=6, 5, 6: number analyzed (Participants) | 6 | 5 | 6
  AUC (0-24), n=6, 5, 6 | 1410 (292.51) | 4940 (1131.6) | 8330 (3363.3)
  AUC (0-168), n=6, 5, 6: number analyzed (Participants) | 6 | 5 | 6
  AUC (0-168), n=6, 5, 6 | 1420 (291.72) | 5080 (1332.6) | 8480 (3249.8)
  AUC (0-inf), n=6, 5, 6: number analyzed (Participants) | 6 | 5 | 6
  AUC (0-inf), n=6, 5, 6 | 1420 (291.72) | 5080 (1328.9) | 8480 (3249.8)

25. Primary Outcome: Cmax, C24 and C168 of GSK3389404 Following Single Dose on Day 1 of Part 2
Description: Blood samples were collected to evaluate Cmax, C24 and C168 of GSK3389404 on Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 15 post-dose.
Time Frame: Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 15 post-dose
Population: Pharmacokinetic Concentration Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  Cmax | 236 (64.551) | 723 (216.01) | 1280 (633.56)
  C24 | 0.00 (0.0000) | 2.58 (6.3278) | 16.7 (20.848)
  C168 | 0.00 (0.0000) | 0.00 (0.0000) | 0.00 (0.0000)

26. Primary Outcome: Tmax, T1/2 and Tlag of GSK3389404 Following Single Dose on Day 1 of Part 2
Description: Blood samples were collected to evaluate Tmax, T1/2 and Tlag of GSK3389404 on Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 15 post-dose.
Time Frame: Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 15 post-dose
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6
Hour
  Tmax, n=6, 6, 6 | 2.33 (1.03) | 2.01 (0.02) | 2.42 (0.92)
  T1/2, n=6, 5, 6: number analyzed (Participants) | 6 | 5 | 6
  T1/2, n=6, 5, 6 | 3.14 (1.0621) | 3.47 (1.8907) | 4.04 (1.7867)
  Tlag, n=6, 6, 6 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

27. Primary Outcome: CL/F of GSK3389404 Following Single Dose on Day 1 of Part 2
Description: Blood samples were collected to evaluate CL/F of GSK3389404 on Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 15 post-dose. Only those participants with data available at the specified time points were analyzed.
Time Frame: Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 15 post-dose
Population: Pharmacokinetic Concentration Population
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 5 | 6
Liter per hour | 22.1 (5.9872) | 12.5 (3.4120) | 15.6 (4.7861)

28. Primary Outcome: AUC(0-24) and AUC From Time Zero to the End of the Dosing Interval [AUC(0-tau)] of GSK3389404 Following Dosing on Day 22 of Part 2
Description: Blood samples were collected to evaluate AUC (0-24) and AUC (0-tau) of GSK3389404 on Day 22 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 29, 36, 50, 71 and at Follow-up (Day 113+- 2 days ).
Time Frame: Day 22 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 29, 36, 50, 71 and at Follow-up (Day 115)
Population: Pharmacokinetic Concentration Population
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6
ng*hour/mL
  AUC (0-24) | 1486 (364.92) | 3973 (906.81) | 8918 (3447.7)
  AUC (0-tau) | 1598 (565.02) | 4052 (873.65) | 9047 (3361.3)

29. Primary Outcome: Observed Concentration at the End of the Dosing Interval (Ctau), C24 and Cmax of GSK3389404 Following Dosing on Day 22 of Part 2
Description: Blood samples were collected to evaluate Ctau, C24 and Cmax of GSK3389404 on Day 22 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 29, 36, 50, 71 and at Follow-up (Day 113+- 2 days ).
Time Frame: as for outcome 28
Population: Pharmacokinetic Concentration Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  Ctau | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  C24 | 0.000 (0.0000) | 4.767 (7.4115) | 15.60 (18.278)
  Cmax | 197.7 (39.657) | 614.8 (211.25) | 1257 (799.88)

30. Primary Outcome: Tmax, T1/2 and Tlag of GSK3389404 Following Dosing on Day 22 of Part 2
Description: Blood samples were collected to evaluate Tmax, T1/2 and Tlag of GSK3389404 on Day 22 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 29, 36, 50, 71 and at Follow-up (Day 113+- 2 days).
Time Frame: as for outcome 28
Population: Pharmacokinetic Concentration Population
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6
Hour
  Tmax | 2.17 (0.98) | 2.26 (0.88) | 2.67 (1.03)
  T1/2 | 4.768 (3.2072) | 3.450 (1.6049) | 3.585 (1.2332)
  Tlag | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

31. Primary Outcome: Cl/F of GSK3389404 Following Dosing on Day 22 of Part 2
Description: Blood samples were collected to evaluate Cl/F of GSK3389404 on Day 22 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 29, 36, 50, 71 and at Follow-up (Day 113+- 2 days).
Time Frame: as for outcome 28
Population: Pharmacokinetic Concentration Population
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6
Liter per hour | 20.50 (6.3906) | 15.48 (3.6973) | 14.39 (3.7029)

32. Secondary Outcome: Dose Proportionality of GSK202007 for Dose Range 10 mg - 120 mg After Single Dose Administrations
Description: Results of dose proportionality assessment using power model and analysis of variance (ANOVA) following single dose administariton (Part 1 and Day 1 in Part 2) are presented. Slope estimates and 90% confidence interval are presented for combined data of Day 1 of Part 1 and 2.
Time Frame: Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 30 post-dose; Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 15 post-dose in Part 2.
Population: Pharmacokinetic Concentration Population (combined for Part 1 and 2). Only data available at the specified time points was analyzed. (represented by n=X in the category titles).
Measure: Number (90% Confidence Interval); unit: ratio
Groups:
- GSK3389404 10-120 mg: Participants received a single dose of either 10 mg or 30 mg or 60 mg or 120 mg of GSK3389404 by subcutaneous injection on Day 1 of Part 1 or Part 2.
Arm/Group | GSK3389404 10-120 mg
Number analyzed (Participants) | 41
ratio
  AUC (0-24), n=40: number analyzed (Participants) | 40
  AUC (0-24), n=40 | 1.08 [0.98 to 1.18]
  AUC (0-inf), n=40: number analyzed (Participants) | 40
  AUC (0-inf), n=40 | 1.07 [0.97 to 1.18]
  Cmax, n=41 | 0.975 [0.83 to 1.12]

33. Secondary Outcome: Dose Proportionality of GSK202007 for Dose Range 30 mg - 120 mg After Multiple Dose Administrations
Description: Results of proportionality assessment using power model and ANOVA following multiple doses are presented. Slope estimates and 90% confidence interval are presented for Day 22 of Part 2.
Time Frame: Day 22 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 29, 36, 50, 71 and at Follow-up (Day 115) in Part 2
Population: Pharmacokinetic Concentration Population
Measure: Number (90% Confidence Interval); unit: ratio
Groups:
- GSK3389404 30-120 mg: Participants received a single dose of either 30 mg or 60 mg or 120 mg of GSK3389404 by subcutaneous injection QW for 4 weeks in Part 2.
Arm/Group | GSK3389404 30-120 mg
Number analyzed (Participants) | 18
ratio
  AUC (0-tau) | 1.25 [1.04 to 1.46]
  Cmax | 1.25 [0.96 to 1.55]

34. Secondary Outcome: Accumulation Ratio by AUC (RAUC), by Cmax (RCmax), by C24 (RC24) and by Ctau (RCtau) of GSK3389404 in Part 2
Description: For Part 2, the extent of accumulation of GSK3389404 was evaluated by comparing AUC (0-tau), Cmax, C24 and Ctau on Day 22 to AUC (0-168), Cmax, C24 and C168 on Day 1. For each dose level, a linear mixed effect model was fitted with the log transformed PK parameter as the dependent variable, day as a fixed effect and subject as a random effect.
Time Frame: Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 15 post-dose; Day 22 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 29, 36, 50, 71 and at Follow-up (Day 115)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6
Ratio
  RAUC, n=6, 5, 6: number analyzed (Participants) | 6 | 5 | 6
  RAUC, n=6, 5, 6 | 1.115 (0.24879) | 0.8596 (0.099034) | 1.094 (0.24035)
  RCmax, n=6, 6, 6 | 0.8683 (0.16676) | 0.8518 (0.18537) | 0.9920 (0.32054)
  RC24, n=0, 1, 3: number analyzed (Participants) | 0 | 1 | 3
  RC24, n=0, 1, 3 |  | 0.8580 (NA) — Only one participant was analyzed at this endpoint, hence standard deviation could not be calculated. | 0.5890 (0.51139)
  RCtau, n=0, 0, 0: number analyzed (Participants) | 0 | 0 | 0

35. Secondary Outcome: Time Invariance (LI) of GSK3389404 in Part 2
Description: For Part 2, time invariance was evaluated by comparing AUC (0-tau) for Day 22 to AUC (0-inf) for Day 1. For each dose level, a linear mixed effect model was fitted with the log transformed PK parameter as the dependent variable, day as a fixed effect and subject as a random effect. Only those participants with data available at the specified time points were analyzed.
Time Frame: as for outcome 34
Population: Pharmacokinetic Concentration Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 5 | 6
Ratio | 1.115 (0.24879) | 0.8598 (0.098644) | 1.094 (0.24035)

36. Secondary Outcome: Trough Plasma Concentrations of GSK3389404 in Part 2
Description: For Part 2, mean plasma GSK3389404 pre-dose values between Day 1 to Day 29 and Ctau were plotted against time to assess attainment of GSK3389404 steady state following multiple dose administration. Achievement of plasma GSK3389404 steady-state was assessed by calculating the 90% confidence interval (CI) of the slope of the linear regression of log (Ctau) versus time. NA indicates data was not available.
Time Frame: Pre-dose on Days 8, 15, 22 and 29
Population: Pharmacokinetic Concentration Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 6 | 6 | 6
Ratio
  Day 8 | NA (NA) — Trough plasma concentrations were below limit of quantification, hence data was not available. | NA (NA) — Trough plasma concentrations were below limit of quantification, hence data was not available. | NA (NA) — Trough plasma concentrations were below limit of quantification, hence data was not available.
  Day 15 | NA (NA) — Trough plasma concentrations were below limit of quantification, hence data was not available. | NA (NA) — Trough plasma concentrations were below limit of quantification, hence data was not available. | NA (NA) — Trough plasma concentrations were below limit of quantification, hence data was not available.
  Day 22 | NA (NA) — Trough plasma concentrations were below limit of quantification, hence data was not available. | NA (NA) — Trough plasma concentrations were below limit of quantification, hence data was not available. | NA (NA) — Trough plasma concentrations were below limit of quantification, hence data was not available.
  Day 29 | NA (NA) — Trough plasma concentrations were below limit of quantification, hence data was not available. | NA (NA) — Trough plasma concentrations were below limit of quantification, hence data was not available. | NA (NA) — Trough plasma concentrations were below limit of quantification, hence data was not available.

37. Secondary Outcome: AUC (0-inf), AUC(0-t), AUC(0-24) of the Metabolite of GSK3389404 After Single Dose in Part 1
Description: Blood samples were collected to evaluate AUC (0-inf), AUC (0-t) and AUC (0-24) of metabolite of GSK3389404 on Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 30 post-dose.
Time Frame: Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 30 post-dose
Population: Pharmacokinetic Concentration Population. Based on emerging PK results during the course of the study, it was observed that metabolite plasma concentrations were not quantifiable in any PK sample. Hence, PK parameters could not be estimated for metabolite.
Arm/Group | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

38. Secondary Outcome: Cmax, C24 and C168 of the Metabolite of GSK3389404 Following Single Dose in Part 1
Description: Blood samples were collected to evaluate Cmax, C24 and C168 of the metabolite of GSK3389404 on Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 30 post-dose.
Time Frame: Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 30 post-dose
Population: as for outcome 37
Arm/Group | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

39. Secondary Outcome: Tmax, T1/2 and Tlag of the Metabolite of GSK3389404 Following Single Dose in Part 1
Description: Blood samples were collected to evaluate Tmax, T1/2 and Tlag of the metabolite of GSK3389404 on Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 30 post-dose.
Time Frame: Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 30 post-dose
Population: as for outcome 37
Arm/Group | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

40. Secondary Outcome: AUC (0-t), AUC(0-24), AUC(0-168) and AUC (0-inf) of the Metabolite of GSK3389404 Following Single Dose on Day 1 of Part 2
Description: Blood samples were collected to evaluate AUC (0-t), AUC (0-24), AUC (0-168) and AUC (0-inf) of the metabolite of GSK3389404 on Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 15 post-dose.
Time Frame: Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 15 post-dose
Population: as for outcome 37
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 0 | 0 | 0

41. Secondary Outcome: Cmax, C24 and C168 of the Metabolite of GSK3389404 Following Single Dose on Day 1 of Part 2
Description: Blood samples were collected to evaluate Cmax, C24 and C168 of the metabolite of GSK3389404 on Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 15 post-dose.
Time Frame: Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 15 post-dose
Population: as for outcome 37
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 0 | 0 | 0

42. Secondary Outcome: Tmax, T1/2 and Tlag of the Metabolite of GSK3389404 Following Single Dose on Day 1 of Part 2
Description: Blood samples were collected to evaluate Tmax, T1/2 and Tlag of the metabolite of GSK3389404 on Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 15 post-dose.
Time Frame: Day 1 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 8 and 15 post-dose
Population: as for outcome 37
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 0 | 0 | 0

43. Secondary Outcome: AUC(0-24) and AUC(0-tau) of the Metabolite of GSK3389404 Following Dosing of GSK3389404 on Day 22 of Part 2
Description: Blood samples were collected to evaluate AUC (0-24) and AUC (0-tau) of the metabolite of GSK3389404 on Day 22 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 29, 36, 50, 71 and at Follow-up (Day 113+- 2 days).
Time Frame: as for outcome 28
Population: as for outcome 37
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 0 | 0 | 0

44. Secondary Outcome: Ctau, C24 and Cmax of the Metabolite of GSK3389404 Following Dosing of GSK3389404 on Day 22 of Part 2
Description: Blood samples were collected to evaluate Ctau, C24 and Cmax of the metabolite of GSK3389404 on Day 22 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 29, 36, 50, 71 and at Follow-up (Day 113+- 2 days).
Time Frame: as for outcome 28
Population: as for outcome 37
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 0 | 0 | 0

45. Secondary Outcome: Tmax, T1/2 and Tlag of the Metabolite of GSK3389404 Following Dosing on Day 22 of Part 2
Description: Blood samples were collected to evaluate Tmax, T1/2 and Tlag of the metabolite of GSK3389404 on Day 22 (pre-dose) and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose; and on Days 29, 36, 50, 71 and at Follow-up (Day 113+- 2 days).
Time Frame: as for outcome 28
Population: as for outcome 37
Arm/Group | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from start of the study treatment up to 62 days in Part 1 and up to 115 days in Part 2.
Description: On treatment SAEs and non-serious AEs were reported for the Safety Population.
Arm/Group | Part 1: Placebo | Part 1: GSK3389404 10 mg | Part 1: GSK3389404 30 mg | Part 1: GSK3389404 60 mg | Part 1: GSK3389404 120 mg | Part 2: Placebo | Part 2: GSK3389404 30 mg | Part 2: GSK3389404 60 mg | Part 2: GSK3389404 120 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/8 | 3/6 | 2/6 | 3/6 | 5/6 | 3/6 | 5/6 | 2/6 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=8) | Part 1: GSK3389404 10 mg (N=6) | Part 1: GSK3389404 30 mg (N=6) | Part 1: GSK3389404 60 mg (N=6) | Part 1: GSK3389404 120 mg (N=6) | Part 2: Placebo (N=6) | Part 2: GSK3389404 30 mg (N=6) | Part 2: GSK3389404 60 mg (N=6) | Part 2: GSK3389404 120 mg (N=6)
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 2
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 2 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.